CLINICAL TRIAL: NCT03201978
Title: A Randomized, Double-Blind, Vehicle-Controlled, 3-Period, Sequential Study to Evaluate Pharmacokinetics, Safety and Tolerability of Single and Repeat Topical Applications of GSK2894512 Cream in Healthy Adult Participants
Brief Title: A Study to Evaluate Pharmacokinetic (PK), Safety and Tolerability of GSK2894512 in Healthy Adult Subjects
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The whole project was discontinued within GSK, hence this study was cancelled before enrolment.
Sponsor: GlaxoSmithKline (Industry)
Collaborators: iCardiac Technologies, Inc. (Industry); Innovaderm Research Inc. (Other); PPD Development, LP (Industry); Algorithme (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 207539
Record Dates: First submitted 2017-06-27; First posted 2017-06-28 (Actual); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Psoriasis
Keywords: Healthy adults; GSK2894512; Topical; Psoriasis; Pharmacokinetics
MeSH Terms: conditions — Psoriasis | interventions — tapinarof

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GSK2894512 cream group (Experimental): Subjects will receive once daily topical repeated application on approximately 5000 cm^2 intact non-occluded skin for 21 days in period 1 followed by once daily on 5000 cm^2 intact occluded skin for 21 days in period 2 (after approximately 21 days of washout period), followed by a single topical application on up to 400 cm^2 gently tape stripped skin area in period 3.
  Interventions: Drug: GSK2894512 1% CREAM
- Vehicle cream group (Placebo Comparator): Subjects will receive once daily topical repeated application on approximately 5000 cm^2 intact non-occluded skin for 21 days in period 1 followed by once daily on 5000 cm^2 intact occluded skin for 21 days in period 2 (after approximately 21 days of washout period), followed by a single topical application on up to 400 cm^2 gently tape stripped skin area in period 3.
  Interventions: Drug: GSK2894512 MATCHING VEHICLE CREAM

INTERVENTIONS:
Drug: GSK2894512 1% CREAM — It will be prepared as close as possible to the time of administration to avoid a prolonged exposure to light. Each single cream application will be made by weight, dispensed on hand (fingertips) covered with clean disposable glove and evenly spread using fingertips.
  Arms: GSK2894512 cream group
Drug: GSK2894512 MATCHING VEHICLE CREAM — It will be prepared as close as possible to the time of administration to avoid a prolonged exposure to light. Each single cream application will be made by weight, dispensed on hand (fingertips) covered with clean disposable glove and evenly spread using fingertips.
  Arms: Vehicle cream group

SUMMARY:
GSK2894512 (trans-isomer) is a fully synthetic, non-steroidal anti-inflammatory agent. This study is being conducted to evaluate the PK, safety and tolerability of GSK2894512 cream, 1 percent administered topically to healthy adult subjects. PK parameters obtained in this study will be used to support the design of future maximum use PK (MUPK) studies in subjects with atopic dermatitis (AD) and plaque psoriasis or psoriasis (PSO). This is a phase 1, randomized, double-blind, vehicle-controlled, 3-period, sequential, inpatient study consists of a Screening visit, 3 treatment periods and a follow-up visit. GSK2894512 cream, 1 percent (or matching vehicle) will be administered sequentially in the treatment periods. Period 1 will include once daily repeated topical applications on approximately 5000 centimeter (cm) ^2 intact non-occluded skin area for 21 days. Period 2 will include once daily repeated topical applications on approximately 5000 cm^2 intact occluded skin area for 21 days. Period 3 will include a single topical application on up to 400 cm^2 gently taped-stripped skin area. Each treatment regimen will be followed by washout period for approximately 21 days, except for Treatment Period 3. Approximately 26 healthy adult subjects will be enrolled in to the study. Total duration of participation in this study will be approximately 18 weeks.

ELIGIBILITY:
* Male or female subjects 18 to 60 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by the investigator on the basis of screening evaluations, including medical history, physical examination, and laboratory tests.
* Body mass index (BMI) within the range of 18 to 30 kilograms (Kg) per meter (m)^2 and body weight >=50 kg. BMI is calculated by taking the subject's weight, in kilograms, divided by the square of the subject's average height, in meters, at screening (BMI = weight in kg divided by height in m^2).
* Non- or ex-smokers; an ex-smoker being defined as someone who completely stopped smoking for at least 6 months before day 1 of this study; the current non-smoking status will be confirmed by urinary cotinine levels.
* A female subject is eligible to participate if she is not pregnant (as confirmed by a negative serum human chorionic gonadotrophin (hCG) test at screening phase between days -29 and -14 and negative serum or urine hCG test on Day -1 prior to each treatment period), not lactating, and at least one of the following conditions applies:

  * not a woman of childbearing potential (WOCBP), or
  * is a WOCBP who agrees to follow the specified contraceptive guidance throughout the study, beginning at least 30 days prior to the first cream application and for at least 30 days after the last cream application of the study.
* Male subject with female partner of childbearing potential must use a male condom and the female partner should use one of the highly effective methods of contraception from the time of first dose of study medication until 30 days after the last cream application of the study.
* Willing to participate and capable of giving signed informed consent.

Exclusion Criteria:

* A history of ongoing serious illness or medical, physical, or psychiatric condition(s) that, in the investigator's opinion, may interfere with the subject's completion of the study.
* A history or presence of skin disorders (e.g., irritant contact dermatitis); history or presence of hypertrophic scarring tissue or keloid formation in scars or needle puncture sites; a tattoo, body piercing or branding located on the study medication application site; excessive body hair that in the Investigator's opinion, may interfere with the areas designated for study medication application.
* Presence or history of AD or PSO.
* Presence of erosions, lacerations, abrasions, dermatitis or any other lesion on the lower legs that could increase absorption of GSK2894512.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Subject has a history of hyperhidrosis.
* Subject had a major surgery within 8 weeks prior to Baseline (Day -1) or has a major surgery planned during the study.
* Known hypersensitivity to GSK2894512 or excipients of the study treatments, or a history of drug or other allergy that, in the opinion of the investigator, contraindicates participation.
* Abnormal aspartate aminotransferase (AST), alanine aminotransferase (ALT) or bilirubin values at screening
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C virus (HCV) antibody and human immunodeficiency virus (HIV) antibody test results at screening.
* Presence of out-of-range cardiac interval (PR <110 millisecond (msec), PR >220 msec, QRS <60msec, QRS >119msec and QTcF > 450msec) on the screening ECG (average of the triplicate ECG) or other clinically significant ECG abnormalities.
* Any history of latent or active tuberculosis (TB) and/or prophylaxis for tuberculosis according to the TB Medical History screening questionnaire.
* Subjects who took an investigational product (in another clinical trial) in the previous 30 days before day 1 of this study.
* Use of any medicated topical product on the same areas as study medication applications within 2 weeks prior to admission to clinical research center (CRC) on Day -1 and throughout each inpatient treatment period.
* Use of any topical products (apart from medicated topical products), except soap and gentle cleansers (example, moisturizers), on the same areas as study medication applications within 2 days prior to admission to CRC on Day -1 and throughout each inpatient treatment period.
* Positive findings of urine drug screen (example, amphetamine, barbiturates, benzodiazepines, cocaine, cannabinoids, opiates, and phencyclidine [PCP]).
* Maintenance therapy with any drug or significant history of drug dependency or alcohol abuse (>3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
* Subjects who have already participated in this clinical study.
* Subjects who donated 50 milliliter (mL) or more of blood in the previous 30 days before day 1 of this study. Donation of 500 mL or more of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc.) in the previous 60 days before Day 1 of this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-14 (Estimated); Primary Completion 2018-05-15 (Estimated); Study Completion 2018-05-15 (Estimated)

PRIMARY OUTCOMES:
Plasma concentrations of GSK2894512 (trans-isomer) | Days 1, 7, 14, 21: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16 hours; Days 2, 3, 8, 9, 15, 16, 22, 23: Pre-dose, in Period-1 and 2. Period-3: Day 1: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 48 hours
  Blood samples will be collected at the indicated time points to evaluate plasma concentration of GSK2894512 (trans-isomer).
Area under the plasma concentration-time curve from time zero to the end of the dosing interval (AUC [0-tau]) of GSK2894512 | Days 1, 7, 14, 21: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16 hours; Days 2, 3, 8, 9, 15, 16, 22, 23: Pre-dose, in Period-1 and 2. Period-3: Day 1: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 48 hours
  Blood sample will be collected at the indicated time points to evaluate PK profile of GSK2894512.
Area under the plasma concentration-time curve from time zero to the last measurable concentration (AUC [0-t) of GSK2894512 | Days 1, 7, 14, 21: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16 hours; Days 2, 3, 8, 9, 15, 16, 22, 23: Pre-dose, in Period-1 and 2. Period-3: Day 1: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 48 hours
  Blood sample will be collected at the indicated time points to evaluate PK profile of GSK2894512.
Maximum observed serum concentration (Cmax) of GSK2894512 | Days 1, 7, 14, 21: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16 hours; Days 2, 3, 8, 9, 15, 16, 22, 23: Pre-dose, in Period-1 and 2. Period-3: Day 1: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 48 hours
  Blood sample will be collected at the indicated time points to evaluate PK profile of GSK2894512.
Time of maximum concentration observed (tmax) of GSK2894512 | Days 1, 7, 14, 21: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16 hours; Days 2, 3, 8, 9, 15, 16, 22, 23: Pre-dose, in Period-1 and 2. Period-3: Day 1: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 48 hours
  Blood sample will be collected at the indicated time points to evaluate PK profile of GSK2894512.
Apparent terminal phase half life (t1/2) of GSK2894512 | Days 1, 7, 14, 21: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16 hours; Days 2, 3, 8, 9, 15, 16, 22, 23: Pre-dose, in Period-1 and 2. Period-3: Day 1: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 48 hours
  Blood sample will be collected at the indicated time points to evaluate PK profile of GSK2894512.
Trough concentration at the end of the dosing interval (Ctau) of GSK2894512 | Days 1, 7, 14, 21: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16 hours; Days 2, 3, 8, 9, 15, 16, 22, 23: Pre-dose, in Period-1 and 2. Period-3: Day 1: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 48 hours
  Blood sample will be collected at the indicated time points to evaluate PK profile of GSK2894512.
Accumulation ratio (Ro) of GSK2894512 | Days 1, 7, 14, 21: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16 hours; Days 2, 3, 8, 9, 15, 16, 22, 23: Pre-dose, in Period-1 and 2. Period-3: Day 1: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 48 hours
  Blood sample will be collected at the indicated time points to evaluate PK profile of GSK2894512.

SECONDARY OUTCOMES:
Number of subjects with any adverse events (AEs) and serious AEs (SAEs) | Up to 14 weeks
  An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other important medical events judged by physician that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the subject or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition.
Number of subjects with abnormal vital sign findings | Up to 13 weeks
  Vital sign parameters including systolic and diastolic blood pressure, heart rate (HR) and body temperature will be evaluated. Vital sign measurements will be preceded by at least 5 minutes of rest (supine or seated) for the subject in a quiet setting.
Number of subjects with abnormal electrocardiogram (ECG) findings | Up to 13 weeks
  Triplicate 12-lead ECG will be obtained using an ECG machine that automatically calculates the HR and measures PR, QRS, QT, and QT interval corrected for heart rate according to Fridericia's formula (QTcF) intervals on Days -1, 3, 9, 16 and 23 in Period-1 and 2; and on Days -1 and 3 in Period-3.
Number of subjects with abnormal findings in digital holter monitoring | Up to 13 weeks
  Continuous digital 12-lead ECGs will be recorded using 12-lead Holter/12-lead ECG recorder from 1 hour prior to dosing to 24 hours after dosing on Days 1, 2, 7, 8, 14, 15, 21 and 22 in period-1 and 2; and on Days 1 and 2 in Period-3.
Number of subjects with abnormal findings in physical examination | Up to 13 weeks
  Complete physical examination will include review of head and neck, heart, lungs, abdomen, skin, general appearance, height and weight.
Number of subjects with abnormal clinical laboratory findings | Up to 13 weeks
  Serum chemistry, hematological and urine analysis parameters will be evaluated.
Assessment of degree of local irritation as a measure of local tolerability | Up to 14 weeks
  Dermal reactions like erythema, edema, papules at test sites will be visually assessed. Degree of local irritation will be assessed to determine tolerability of topical application of GSK2894512 cream. if a subject is found to meet a dermal response graded 4 (definite edema) and above indicated in Erythema and Dermal Response Grading Scale, the study medication applications will be discontinued. Grade <4 will be recorded as an AE.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline